CLINICAL TRIAL: NCT05771376
Title: The Effects of Baduanjin Qigong Exercise Via Telerehabilitation in Ankylosing Spondylitis: A Randomized Controlled Study
Brief Title: The Effects of Baduanjin Qigong Exercise on Ankylosing Spondylitis: A Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Gokce Yagmur Gunes Gencer, Associate Professor, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Qigong Exercise in AS
Record Dates: First submitted 2023-03-05; First posted 2023-03-16 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Ankylosing Spondylitis
Keywords: Qigong Exercises; Ankylosing Spondylitis; Pain; Quality of Life; Fatigue
MeSH Terms: conditions — Spondylitis, Ankylosing; Pain; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients who performed the Qigong exercise program
  Interventions: Other: Qigong exercise program
- Control Group (Experimental): Patients who performed a home exercise program
  Interventions: Other: Home exercise program

INTERVENTIONS:
Other: Qigong exercise program — The intervention group will perform a qigong exercise program online (via Zoom video conference) for 12 weeks under the supervision of two physiotherapists. The qigong exercise program had previously been videotaped by the researchers.
  qigong exercise program includes: Preparation posture Prop up the sky by two improve trijiao Draw a bow on both sides like shooting a vulture Raise single arm up to regulate spleen Look back to treat five strains and seven impairments Shake the head and wag to expel Heart (Xin)-fire Pull toes with both hands to reinforce the kidney Clench one's fist and glare to increase strength Rise and fall on tiptoe sevan times to treat all diseases Ending posture. Qigong exercises will be performed 45 minutes twice in a week for 12 weeks.
  Arms: Intervention Group
Other: Home exercise program — The home exercise program will include stretching for cervical, thoracic and lumbar flexibility, shoulder girdle, hamstring and erector spinal muscles, and strengthening exercises for abdominal, back, and proximal muscles.
  Home exercises will be performed 45 minutes twice in a week for 12 weeks.
  Arms: Control Group

SUMMARY:
The aim of this study is to examine the effectiveness of 12-week Baduanjin qigong exercises in patients with ankylosing spondylitis. 59 volunteer individuals, ages 18-64, will be included in the study. They will be randomly divided into two groups (the intervention and the control). The intervention group will perform a qigong exercise program online (via Zoom video conference) for 12 weeks under the supervision of two physiotherapists. The qigong exercise program had previously been videotaped by the researchers. The control group will perform the home exercise program at home for 12 weeks.

DETAILED DESCRIPTION:
This study will be conducted to examine the effect of Baduanjin qigong exercises on patients with ankylosing spondylitis. 29 individuals with ankylosing spondylitis (the intervention group) and 30 healthy individuals (the control group), totaling 59 volunteer individuals ages 18-64, will be included in the study.

The intervention group will perform a qigong exercise program online (via Zoom video conference) for 12 weeks under the supervision of two physiotherapists. The qigong exercise program had previously been videotaped by the researchers. The control group will perform the home exercise program at home for 12 weeks. The intervention group will perform Qigong online exercise program, and the control group will perform home exercises for 45 minutes twice a week for 12 weeks.

In this study the Bath Ankylosing Spondylitis Disease Activity Index, Bath Ankylosing Spondylitis Functional Index, Bath Ankylosing Spondylitis Metrology Index, Chest Expansion Measurement, The Pittsburgh Sleep Quality Index, Fatigue Severity Scale, Hospital Anxiety and Depression Scale, and Ankylosing Spondylitis Quality of Life Questionnaire will be applied before and after the 12-week exercise program in the evaluation of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ankylosing spondylitis diagnosis

Exclusion Criteria:

* Patients with another rheumatological diseases or orthopedic, neurological, psychiatric, cardiovascular, oncological comorbidities

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2022-02-13 (Actual); Primary Completion 2023-01-07 (Actual); Study Completion 2023-04-07 (Actual)

PRIMARY OUTCOMES:
Disease activity | 12 weeks
  The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) will be used to assess disease activity. The index, designed by a multidisciplinary team with input from patients, consists of six 10 cm horizontal visual analog scales to measure severity of fatigue, spinal and peripheral joint pain, localized tenderness and morning stiffness (both qualitative and quantitative). The final BASDAI score has a range of 0 to 10.
Functional capacity | 12 weeks
  The functional capacity of the patient will be evaluated with The Bath Ankylosing Spondylitis Functional Index (BASFI). BASFI is a set of 10 questions designed to determine the degree of functional limitation in patients with Ankylosing Spondylitis (AS). The 10 questions were chosen with a major input from patients with AS. The first 8 questions are about everyday tasks and dependent on functional anatomy (bending, reaching, changing position, standing, turning, and climbing steps with or without rail) while the final 2 questions assess the patients' ability to cope with everyday life. Each item is scored on a scale of 0-10.
Axial involvement | 12 weeks
  Axial involvement in the patient will be evaluated with the Bath Ankylosing Spondylitis Metrology Index. The Bath AS Metrology Index (BASMI) is a validated composite index of spinal and hip mobility comprising measures of cervical rotation, tragus-to-wall distance, lumbar spinal forward and side flexion, and hip abduction.
Sleep Quality | 12 weeks
  The Pittsburgh Sleep Quality Index will be used to evaluate the sleep quality of patients. The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval.
Fatigue | 12 weeks
  Fatigue Severity Scale (FSS) will be used to evaluate patients' fatigue levels. Fatigue is an overwhelming sense of tiredness and lack of energy that can impair participation in daily tasks and work. It may become a chronic and disabling problem in daily life of the patients with Ankylosing Spondylitis. The FSS is a measurement of fatigue impact on functioning.
Chest expansion | 12 weeks
  Chest expansion will be evaluated by chest expansion measurement. After measuring the chest circumference following a deep inspiration from the fourth intercostal space (at the level of the nipples), chest expansion is determined by measuring again after a forced expiration and taking the net difference between them. The average of two the correct measurements will be taken as the final measurement.
Ankylosing Spondylitis Quality of Life | 12 weeks
  Ankylosing Spondylitis Quality of Life Questionnaire-ASQoL will be used to evaluate the patient's quality of life. ASQoL questionnaire measures disease-specific quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Gokce Yagmur Gunes Gencer, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No